CLINICAL TRIAL: NCT02668848
Title: The Fluid Therapy Strategy of the Patients With Acute Ischemic Stroke and a Bun/Cr Ratio Less Than 15.
Brief Title: The Fluid Therapy Strategy of the Non-dehydrated Patients With Acute Ischemic Stroke.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMRPG6e0401
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2016-07

CONDITIONS: Stroke; Dehydration
Keywords: Stroke; Dehydration; Fluid therapy
MeSH Terms: conditions — Stroke; Dehydration | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- urine monitoring group (Experimental): Patients of urine monitoring group will be checked for urine specific gravity (USG) once between 6a.m. to 12 m.d. in the first 5 days after admission. Patients will be advised to have water according to the level of USG.
  Interventions: Dietary Supplement: water

INTERVENTIONS:
Dietary Supplement: water — If USG>1.02, patients will be advised to drink water via oral or tubal feeding with a dose of 5cc/kg body weight , maximum 300cc, and repeat the same amount of water after dinner in the same day.

SUMMARY:
The investigators previously found that a blood urea nitrogen/creatinine (BUN/Cr) ratio >15 is an independent predictor of early deterioration after acute ischemic stroke. Another study was conducted to determine whether urine specific gravity, another indicator of hydration status and one more easily obtained, is also an independent predictor of early deterioration or stroke-in-evolution (SIE) in such patients. The investigators also conducted a preliminary study, enrolling ischemic stroke patients with a BUN/Cr ratio >15 and find daily Bun/Cr based hydration help to decrease post stroke infection rate and improve 3 months functional outcome. In this study, daily urine specific gravity will be used to adjust hydration therapy in ischemic stroke patients with initial Bun/Cr ratio <15. The primary outcome is the post stroke infection rate in the first 7 days after admission, and secondary outcome is 3 months functional outcome using mRS.

DETAILED DESCRIPTION:
Stroke remains a major medical issue. According to the American Heart Association (AHA) report in 2012, a new or recurrent stroke occurs in around 795,000 people each year, and 1 out of every 18 deaths in the United States is due to stroke. The incidence of stroke may be even higher in the Chinese population than in the US population. In Taiwan, the average annual incidence rate of first-ever stroke for people above 36 years is 330 per 100,000. The associated disease burden of stroke is increasing annually and remains a significant health concern. Common medical complications of stroke include infections, falls, pressure sores, and depression. A systematic review showed that 30% of patients develop post-stroke infection. Though rates of pneumonia and urinary tract infection after stroke are both 10%, pneumonia is associated with higher mortality. If stroke patients become infected during admission, they may experience neurologic deterioration, poor functional outcome, and increased length of stay (LOS).

Adequate hydration is necessary for maintenance of physiologic homeostasis. Dehydration is a frequent cause of mortality in elderly patients. Dehydration is a common and early feature of acute ischemic stroke and may be a contributor to poor outcomes. In the absence of known biological markers of dehydration, biochemical data were analyzed to identify such markers. These studies showed that the blood urea nitrogen (BUN)/creatinine (Cr) ratio ≥ 15 can be used as a marker of dehydration. Our previous study also revealed that BUN/Cr ratio ≥ 15 is an independent predictor of stroke-in-evolution (SIE). These studies suggest that BUN/Cr ratio may used to identify those patients with acute ischemic stroke who are dehydrated and will benefit from hydration therapy.

The investigators then conducted a phase II single arm control trial of patients with acute ischemic stroke and BUN/Cr ratio ≥15 conducted from January 2011 to December 2013. The results demonstrated blood urea nitrogen/creatinine (BUN/Cr)-based hydration therapy decreases the length of stay (LOS) and rate of post-stroke infection.

Since the BUN/Cr ratio is an indicator of hydration status, and urine specific gravity is also an indicator of hydration status, the investigators hypothesized that urine specific gravity would also be an independent predictor of early deterioration. A urine specific gravity >1.010 indicates that urine is concentrating in the kidneys which means that the body might be relatively dehydrated. Because such an increase in urine specific gravity occurs earlier than an increase in the BUN/Cr ratio, the investigators thought that an increase in urine specific gravity might be an earlier predictor of early deterioration in ischemic stroke than the BUN/Cr ratio.

In this study, daily urine specific gravity will be used to adjust hydration therapy in ischemic stroke patients with initial Bun/Cr ratio <15. The primary outcome is the post stroke infection rate in the first 7 days after admission, and secondary outcome is 3 months functional outcome using mRS.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke diagnosed by the clinical presentations and brain imaging is confirmed by a stroke care specialist,
2. has a measurable neurologic deficit according to the National Institutes of Health Stroke Scale (NIHSS),
3. the time between the onset of neurological symptoms and starting therapy are less than 48 hours,
4. admission BUN/Cr<15

Exclusion Criteria:

1. no informed consent obtained,
2. initial NIHSS >15,
3. prepared for or received fibrinolytic therapy,
4. prepared for or received surgical intervention with 14 days,
5. congestive heart failure according to past history or Framingham criteria,
6. history of liver cirrhosis or severe liver dysfunction (ALT or AST > x 3 upper normal limit),
7. admission blood Cr >2 mg/dl,
8. initial blood pressure SBP<90 mmHg,
9. fever with core temperature >=38°C,
10. indication of diuretics for fluid overload,
11. any conditions needed more aggressive hydration or blood transfusion,
12. cancer under treatment,
13. life expectancy or any reasons for follow-up < 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
the rate of post-stroke infection | the first 7 days after admission
  The post-stroke infection is defined as a core body temperature>38C in any time point.

SECONDARY OUTCOMES:
functional outcome | 3 months after ischemic stroke
  We use modified Rankin scale for neurological evaluation to assess whether USG based hydration therapy results in clinical benefit at three months.

CONTACTS AND LOCATIONS:
Overall Officials: Leng C Lin, M.D., Principal Investigator — Department of Emergency Medicine, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lin LC, Lee JD, Hung YC, Chang CH, Yang JT. Bun/creatinine ratio-based hydration for preventing stroke-in-evolution after acute ischemic stroke. Am J Emerg Med. 2014 Jul;32(7):709-12. doi: 10.1016/j.ajem.2014.03.045. Epub 2014 Apr 4. PMID 24768671
- [Result] Lin WC, Shih HM, Lin LC. Preliminary Prospective Study to Assess the Effect of Early Blood Urea Nitrogen/Creatinine Ratio-Based Hydration Therapy on Poststroke Infection Rate and Length of Stay in Acute Ischemic Stroke. J Stroke Cerebrovasc Dis. 2015 Dec;24(12):2720-7. doi: 10.1016/j.jstrokecerebrovasdis.2015.08.002. Epub 2015 Aug 31. PMID 26338107